CLINICAL TRIAL: NCT01339624
Title: Nasal Fentanyl And Renal Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: MASSIMILIANO ETTERI, VALDUCE HOSPITAL
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NASAL FENTANYL-01
Record Dates: First submitted 2011-04-15; First posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2009-09

CONDITIONS: Acute Renal Colic
Keywords: analgesia; renal colic; ketorolac; nasal fentanyl; morphine.; treatment of acute renal colic
MeSH Terms: conditions — Renal Colic; Agnosia | interventions — Fentanyl; Ketorolac Tromethamine; Morphine

ARMS (2):
- NASAL FENTANYL, (Active Comparator)
  Interventions: Drug: FENTANYL
- KETOROLAC + MORPHINE (Active Comparator)
  Interventions: Drug: Ketorolac Tromethamine AND morphine

INTERVENTIONS:
Drug: FENTANYL — FENTANYL CITRATE, NASAL, 3 GAMMA/KG
  Arms: NASAL FENTANYL,
Drug: Ketorolac Tromethamine AND morphine — morphine 5 MG diluted in saline solution 100 ml followed by 2-ml ampoule of ketorolac 30 MG in saline solution 100 ml was infused:
  Arms: KETOROLAC + MORPHINE

SUMMARY:
The purpose of this study is to determine whether nasal fentanyl is effective in the treatment of renal colic in adults in emergency department.

ELIGIBILITY:
Inclusion Criteria:

* The patients were adults aged 18 to 65 years, presenting in ED with classical clinical symptoms of renal colic (sudden monolateral flank pain with inguinal irradiation) with a 10-cm visual analog scale (VAS) greater than or equal to 7

Exclusion Criteria:

* Were analgesia within 6 hours of arrival
* Allergy to opiates and NSAIDs
* Opiates abuse, known or suspected abdominal aortic dissection or aneurism,
* Presence of peritonitis
* Hemodynamic instability
* Pregnancy, breastfeeding, anticoagulant therapy.
* Patients with known renal, pulmonary, cardiac or hepatic failure, as well as those with renal transplantation, were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in visual analogue scale pain intensity score | 30 and 60 minutes
  This measure was obtained using a 10-cm with marked numbers visual analog scale (VAS score).

SECONDARY OUTCOMES:
Use of rescue therapy at 30 minutes | 30 MINUTES
The occurrence of adverse events | 60 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, Italy